CLINICAL TRIAL: NCT05180162
Title: Imaging of Pathologic Fibrosis Using 68Ga-FAP-2286
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Hope (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Thomas Hope, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-32872
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Liver Fibrosis; Pulmonary Fibrosis; Myocardial Fibrosis
Keywords: Positron Emission Tomography (PET); Imaging; 68Ga-FAP-2286
MeSH Terms: conditions — Liver Cirrhosis; Pulmonary Fibrosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Liver Fibrosis (Experimental): Patients with liver fibrosis will receive a single administration of 68Ga-FAP-2286 prior to PET imaging.
  Interventions: Drug: 68Ga-FAP-2286; Procedure: Positron Emission Tomography (PET)
- Cohort 2: Pulmonary Fibrosis (Experimental): Patients with pulmonary fibrosis will receive a single administration of 68Ga-FAP-2286 prior to PET imaging.
  Interventions: Drug: 68Ga-FAP-2286; Procedure: Positron Emission Tomography (PET)
- Cohort 3: Myocardial Fibrosis (Experimental): Patients with myocardial fibrosis will receive a single administration of 68Ga-FAP-2286 prior to PET imaging.
  Interventions: Drug: 68Ga-FAP-2286; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: 68Ga-FAP-2286 — A dose of 3 - 8 millicurie (mCi) will be given intravenously (IV)
  Other Names: 68Gallium-Fibroblast Activation Protein-2286
Procedure: Positron Emission Tomography (PET) — Imaging will begin 50-100 minutes after injection and last about 45 minutes.
  Other Names: PET Imaging; PET Scan

SUMMARY:
This is a single arm prospective pilot trial that evaluates the ability of a novel imaging agent (68Ga-FAP-2286) to identify pathologic fibrosis in the setting of hepatic, cardiac and pulmonary fibrosis.

FAP-2286 is a peptide that potently and selectively binds to Fibroblast Activation Protein (FAP). FAP is a transmembrane protein expressed on fibroblasts and has been shown to have higher expression in idiopathic pulmonary fibrosis (IPF), cirrhosis, and cardiac fibrosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. All cohorts: Safety of 68Ga-FAP-2286.

II. Cohort 1: Measured uptake of radiotracer (SUVpeak) in regions of known liver fibrosis.

III. Cohort 2: Measured uptake of radiotracer (SUVpeak) in regions of known pulmonary fibrosis.

IV. Cohort 3: Measured uptake of radiotracer (SUVpeak) in regions of myocardial fibrosis.

EXPLORATORY OBJECTIVES:

I. Correlation of 68Ga-FAP-2286 uptake with FAP expression determined by immunohistochemistry.

II. Compare 68Ga-FAP-2286 scan results to archival Computerized tomography (CT), magnetic resonance imaging (MRI), or Positron Emission Tomography (PET) images.

Patients will receive a single administration of 68Ga-FAP-2286 prior to PET imaging and will be followed for up to two hours after the injection of 68Ga-FAP-2286 for evaluation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Confirmed pathologic fibrosis in one of the following cohorts

   1. Cohort 1: Hepatic fibrosis, based on cirrhosis on imaging or hepatic fibrosis on liver biopsy.
   2. Cohort 2: Pulmonary fibrosis, based on CT findings or biopsy of lung parenchyma.
   3. Cohort 3: High likelihood of cardiac fibrosis as indicated by known cardiac sarcoidosis or amyloidosis (shown on MRI or Fluorodeoxyglucose (FDG) PET), recent myocardial infarction within the last 30 days (as shown by an elevated troponin), known cardiotoxicity (decreased ejection fraction on systemic therapy), or other known inflammatory or infiltrative disease.
3. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Unlikely to comply with protocol procedures, restrictions and requirements and judged by the Investigator to be unsuitable for participation.
2. Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with treatment-related adverse events | Up to 31 days
  Proportion of participants with Adverse Events, as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 will be reported.
Median peak standardized uptake value (SUVpeak) in liver region | Up to 1 days
  The median SUVpeak in regions of known liver fibrosis will be reported with 95% confidence intervals
Median peak standardized uptake value (SUVpeak) in lung region | Up to 1 days
  The median SUVpeak in regions of known pulmonary fibrosis will be reported with 95% confidence intervals
Median peak standardized uptake value (SUV) in myocardium region | Up to 1 days
  The median SUVpeak in regions of known myocardial fibrosis will be reported with 95% confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No